CLINICAL TRIAL: NCT06869577
Title: Project SUGRI - a Supportive Group Intervention for Caregivers to Patients Diagnosed With a Glioblastoma
Brief Title: A Supportive Group Intervention for Caregivers to Patients Diagnosed With a Glioblastoma
Acronym: SUGRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other); The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Tiit Mathiesen, Tiit Mathiesen, Professor in Neurosurgery, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Project SUGRI - F-24004933; Copenhagen University Hospital (Other Grant/Funding Number: The Danish Cancer Society:R344-A19341, Novo Nordisk Foundation: NNF22OC0080425)
Record Dates: First submitted 2025-01-03; First posted 2025-03-11 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Caregiver; Glioblastoma Multiform (Grade IV Astrocytoma)
Keywords: caregiver; intervention; group; supportive care; glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A supportive group intervention (Experimental): The intervention consists of following four elements:
  * Weekly HCP facilitated online group meetings for caregivers (n=12) over three months
  * Access to a webpage with informational videos of health care professionals and videos with other caregivers
  * Offer a box of reflection cards and cards to provide caregivers with help
  * Access to a closed online Facebook group
  Interventions: Other: Project SUGRI: A supportive group intervention for caregivers to patients with a glioblastoma

INTERVENTIONS:
Other: Project SUGRI: A supportive group intervention for caregivers to patients with a glioblastoma — A 12-week supportive group intervention targeted caregivers to patients with glioblastoma.

SUMMARY:
Feasibility test and evaluation of a group intervention for caregivers to patients diagnosed with a glioblastoma.

DETAILED DESCRIPTION:
Methods and design:

The study is a three-phase sequential mixed-method feasibility study. The overall framework is guided by the British Medical Research Council framework for developing Complex Intervention. The study will apply Patient and Public Involvement (PPI) to design and develop the intervention. The study will test the feasibility of the newly designed group intervention.

Participants:

Family caregivers (≥18 years) to patients (≥18 years) diagnosed with a GBM grade IV or diffuse astrocytoma grade IV offered standard oncological treatment. Participants must be able to understand, read, and speak Danish.

Intervention:

The intervention runs over 12 weeks. Caregivers are offered weekly online meetings in a group of 12 caregivers facilitated by a HCP. Moreover, they are offered access to a website with 15 videos. 8 videos where HCPs share information knowledge relevant for the disease- and treatment trajectory. And 7 videos where other caregivers sharing their care experiences. The intervention also includes a box of reflection cards, that caregivers are given, when they are included in the intervention. The reflection cards present a question for the caregiver, followed by a quote from a caregiver and knowledge regarding the subject of the card. Caregivers are also invited into a closed online group on FaceBook, where they can write within the group.

Data collection:

Primary outcome is feasibility of the intervention. Secondary outcomes are following reported outcome date at baseline and post-intervention:

Caregivers will complete following three questionnaires: The Caregiver Role and Responsibility Scale (CRRS), to assess broad life impacts for caregiver, the Iceland-Family Perceived Support Questionnaire (ICE-FPSQ) to measures families perceived support from nurses and other healthcare professionals providing the intervention. The Hospital Anxiety and Depression Scale (HADS) to measure symptoms of anxiety and depression.

Patients will complete following three questionnaires: the Functional Assessment of Cancer Therapy - Brain (FACT-Br) to assess the patients' health related QOL, the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) to measure patients' symptom prevalence, intensity, and interference with the daily life. The Hospital Anxiety and Depression Scale (HADS) to measure symptoms of anxiety and depression.

Data will be collected electronically using RedCap. Demographic data of the participants will be completed at baseline and information on patient histology will be obtained from the patient's medical journal and stored in RedCap.

The intervention will also be evaluated qualitatively by individually semi structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers (≥18 years) to patients (≥18 years) diagnosed with a GBM grade IV or diffuse astrocytoma grade IV offered Stupps treatment regime.

Exclusion Criteria:

* Participants who do not understand, read, and speak Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility parametres | The final evaluation of the feasibility of the intervention will be conducted after the completion of the intervention, which is scheduled to last 12 weeks.
  The primary outcome is the feasibility of the intervention. Accurate feasibility parameters will be outlined when the intervention is fully designed. However, we will most likely access recruitment rate, adherence to the overall intervention, acceptability, and safety. We will establish the final percentages for feasibility within each parameter prior test of the intervention and use these to report the overall feasibility of the intervention. Final percentages will be guided by other feasibility studies within the neuro-oncology field.
Feasibility parametres | The final evaluation of the feasibility of the intervention will be conducted after the completion of the intervention, which is scheduled to last 12 weeks.
  Feasibility of the intervention will also be accessed by a survey. We will develop a study specific questionnaire to evaluate the content and overall intervention. The questionnaire will apply a 5-point Likert scale to evaluate the intervention. The questionnaire will be developed when the final intervention is designed.

SECONDARY OUTCOMES:
Quantitative PRO data | Secondary outcomes are PRO data completed by caregivers and patients at baseline, post intervention (12 weeks), and at follow-up (18 weeks)..
  Caregiver outcome 1:
  - The Caregiver Role and Responsibility Scale (CRRS) to assess broad life impacts for caregivers (0-164 POINTS)
Quantitative PRO data | Secondary outcomes are PRO data completed by caregivers and patients at baseline, post intervention (12 weeks), and at follow-up (18 weeks).
  Caregiver outcome 2:
  - The Iceland-Family Perceived Support Questionnaire (ICE-FPSQ) to measures families perceived support from nurses and other healthcare professionals (14-70 POINTS)
Quantitative PRO data | Secondary outcomes are PRO data completed by caregivers and patients at baseline, post intervention (12 weeks), and at follow-up (18 weeks).
  Caregiver outcome 3:
  - The Hospital Anxiety and Depression Scale (HADS) to measure symptoms of anxiety and depression (0-21 POINTS)
Quantitative PRO data | Secondary outcomes are PRO data completed by caregivers and patients at baseline, post intervention (12 weeks), and at follow-up (18 weeks).
  Patient outcomes 1:
  - The Functional Assessment of Cancer Therapy - Brain (FACT-Br) to assess the patients' health related quality of life (0-200 POINTS)
Quantitative PRO data | Secondary outcomes are PRO data completed by caregivers and patients at baseline, post intervention (12 weeks), and at follow-up (18 weeks).
  Patient outcomes 2:
  - The MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) to measure patients' symptom prevalence, intensity, and interference with the daily life (0-220 POINTS)
Quantitative PRO data | Secondary outcomes are PRO data completed by caregivers and patients at baseline, post intervention (12 weeks), and at follow-up (18 weeks).
  Patient outcomes 3:
  - The Hospital Anxiety and Depression Scale (HADS) to measure symptoms of anxiety and depression (0-21 POINTS)
Qualitative interview data | Post-intervention (Week 12)
  Semistructured interviews will be carried out with all caregivers after compleation of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No